CLINICAL TRIAL: NCT02938013
Title: deLIVER: Direct Acting Antiviral Effects on the Liver
Acronym: deLIVER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00110677
Record Dates: First submitted 2016-10-12; First posted 2016-10-19 (Estimated); Results first posted 2020-11-16 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2020-10

CONDITIONS: HCV Coinfection; Liver Disease; HIV
MeSH Terms: conditions — Liver Diseases | interventions — Sofosbuvir; velpatasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Monoinfected: Sofosbuvir/Velpatasvir/Voxilaprevir SOF/VEL/VOX days 0-7 Paired liver biopsy at days 0 and 7 (cohort 1) or days 0 and 4 (cohort 2). SOF/VEL days 8 (week 2) through 84 (week 12). Post-treatment follow up through week 12.
  Interventions: Drug: Sofosbuvir/Velpatasvir/Voxilaprevir [SOF/VEL/VOX]
- Group B (Active Comparator): Monoinfected: Sofosbuvir/Velpatasvir (SOF/VEL) days 0 through 7 and Paired liver biopsy at days 0 and 7 (cohort 1) or days 0 and 4 (cohort 2). SOF/VEL on day 8 (week 2) through 84 (week 12) . Post-Treatment follow up through week 12.
  Interventions: Drug: Sofosbuvir/Velpatasvir (SOF/VEL)
- Group C (Active Comparator): HIV/HCV Co-infection: Sofosbuvir/Velpatasvir (SOF/VEL) days 0 through 7 and Paired liver biopsy at days 0 and 7 (cohort 1) or days 0 and 4 (cohort 2). SOF/VEL on day 8 (week 2) through 84 (week 12) . Post-Treatment follow up through week 12.
  Interventions: Drug: Sofosbuvir/Velpatasvir (SOF/VEL)

INTERVENTIONS:
Drug: Sofosbuvir/Velpatasvir/Voxilaprevir [SOF/VEL/VOX] — antiviral therapy for HCV
  Arms: Group A
Drug: Sofosbuvir/Velpatasvir (SOF/VEL) — antiviral therapy for HCV
  Arms: Group B; Group C

SUMMARY:
Open-label, partially-randomized plasma and liver sampling study to assess hepatitis C virus (HCV) kinetics during treatment with two (Sofosbuvir/Velpatasvir) or three (Sofosbuvir/Velpatasvir/Voxilaprevir) direct acting antivirals (DAAs)

DETAILED DESCRIPTION:
Primary Objective: The primary objective is to estimate the 1-week change in the proportion of HCV-infected hepatocytes in participants with HCV monoinfection and HIV/HCV coinfection on therapy with two or three DAAs with different mechanisms of action using single cell laser microdissection (scLCM).

Secondary Objectives:

Estimate the change over the first week in plasma HCV RNA in subjects with HCV monoinfected and HIV/HCV coinfected participants on therapy with two or three DAAs

Estimate the 1 week change in the amount of HCV RNA per infected hepatocyte using scLCM on liver biopsy specimens, obtained just prior to treatment initiation (pre-treatment), and after the first week of DAA therapy.

Estimate the change in the proportion of HCV-infected hepatocytes that express interferon-stimulated genes (ISGs) within the first week of DAA therapy using scLCM.

Measure the change in expression of ISGs in non-parenchymal intrahepatic immune cells (Kupffer cells, plasmacytoid dendritic cells) within the first week of DAA therapy using scLCM.

Exploratory Objectives:

Estimate the 1 week change in expression of ISGs from peripheral blood mononucleated cells (PBMCs) within the first week of DAA+ribavirin (RBV) therapy using scLCM.

Compare sequence(s) of HCV protease, nonstructural protein 5A (NS5A), and nonstructural protein 5B (NS5B) depending on the peripheral sequence) of intrahepatic HCV RNA in single cells and bulk tissue, before and during week 1 of DAA+RBV therapy.

Estimate the week 1 change in the sizes and numbers of HCV-infected clusters on DAA therapy to test whether clearance of HCV-infected hepatocytes occurs in spatially random patterns or within specific clusters.

ELIGIBILITY:
Inclusion Criteria Participants must meet all of the following inclusion criteria to be eligible for participation

1. Ability and willingness of participant to provide written informed consent.
2. Men and women age ≥18 to ≤70 years at study entry
3. Body mass index (BMI) ≥ 18 kg/m2
4. HCV RNA ≥ 10,000 IU/mL at Screening
5. HCV genotype 1a at Screening or within 6 months of screening
6. Chronic HCV infection (≥ 6 months) documented by prior medical history
7. HCV treatment-naïve with no prior treatment with any IFN, RBV, or approved or experimental HCV-specific DAA
8. Absence of cirrhosis as defined as transient elastography (FibroScan®) liver stiffness measurement < 12.5 kPa within 6 months of screening
9. The following laboratory values obtained within 42 days prior to study entry. • Hemoglobin > 10 g/dL for men and > 9 g/dL for women

   • Platelet count ≥90,000/mm3

   • International normalized ratio (INR) ≤1.5

   • Calculated creatinine clearance (CrCl) ≥ 30 mL/min

   • Alanine aminotransferase (ALT) and aspartate aminotransferase level ≤ 10 x upper limit of the normal range (ULN)

   • Total bilirubin <3 mg/dL

   • Albumin ≥3.5 g/dL
   * CD4+ cell count ≥200 cells/uL and CD4+ cell percentage ≥14% within 42 days of study entry at any US laboratory that has a Clinical Laboratory Improvement Amendments (CLIA) certification [HIV seropositive participants only]
   * HIV RNA < 400 copies/mL prior to study entry by any US laboratory that has a CLIA certification or its equivalent [HIV seropositive participants only]
10. On a qualifying antiretroviral therapy (ART) regimen which is permitted with SOF/VEL. This allows for antiretroviral regimen that does not include Efavirenz, Nevirapine, or Tipranavir.
11. Women of childbearing potential must have a negative serum pregnancy test at Screening and a negative urine pregnancy test on Day 0 prior to liver biopsy
12. All participants must agree not to participate in a conception process (e.g., active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization).
13. If participating in sexual activity that could lead to pregnancy, the participant (men and women) must also agree to use two reliable methods of contraception simultaneously while receiving study treatment and for 30 days after stopping study treatment.

    A combination of TWO of the following contraceptives MUST be used appropriately:

    • Condoms (male or female) with or without a spermicidal agent

    • Diaphragm or cervical cap with spermicide

    • IUD (intrauterine device)
14. Participants who are not of reproductive potential (women who have been post-menopausal for at least 24 consecutive months or have undergone hysterectomy, bilateral tubal ligation, and/or bilateral oophorectomy or men who have documented azoospermia) are eligible without requiring the use of contraceptives. Acceptable documentation of sterilization and menopause is specified below.

    Written or oral documentation communicated by clinician or clinician's staff of one of the following:
    * Physician report/letter
    * Laboratory report of azoospermia
    * Follicle stimulating hormone-release factor (FSH) measurement elevated into the menopausal range as established by the reporting laboratory.
15. Participants must be able to adhere to dosing instructions for study drug administration and able to complete the study schedule of assessments, in the opinion of the investigator.

Exclusion Criteria

Subjects who meet any of the following exclusion criteria are not to be enrolled in this study:

1. Breastfeeding.
2. Known allergy/sensitivity or any hypersensitivity to components of study drugs or their formulation.
3. Acute or serious illness requiring systemic treatment and/or hospitalization within 42 days prior to study entry.
4. Active hepatitis B infection (positive HBsAg) within 42 days prior to study entry.
5. History of decompensated liver disease (including but not limited to encephalopathy, variceal bleeding, or ascites) prior to study entry.
6. Any cause of liver disease other than chronic HCV infection, including but not limited to the following:

   • Hemochromatosis
   * Alpha-1 antitrypsin deficiency
   * Wilson's disease
   * Autoimmune hepatitis
   * Alcoholic liver disease
   * Drug-related liver disease
7. Uncontrolled or active depression or other psychiatric disorder within 24 weeks prior to study entry that in the opinion of the investigator might preclude adherence to study requirements.
8. Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements.
9. Serious illness including uncontrolled seizure disorders, active coronary artery disease within 24 weeks prior to study entry, or other chronic medical conditions that in the opinion of the investigator might preclude completion of the protocol.
10. Presence of active or acute AIDS-defining opportunistic infections within 12 weeks prior to study entry.
11. Active or history of malignancy within 2 years prior to study entry other than basal cell carcinoma of the skin and/or cutaneous Kaposi's sarcoma (KS) and/or cervical or anal dysplasia or carcinoma in situ.

13. Infection with any HCV genotype other than genotype 1a, or mixed genotype infection any time prior to study entry.

14. History of major organ transplantation with an existing functional graft any time prior to study entry.

15. History of acquired or hereditary bleeding disorder (e.g., hemophilia, warfarin use) or any other cause of or tendency toward excessive bleeding time prior to study entry.

16. Gastrointestinal disorder or post-operative condition that could interfere with the absorption of the study drug 17. Difficulty with blood collection and/or poor venous access for the purposes of phlebotomy 18. Planning to take any of the following medications or supplements from Day -7 to the end of treatment:

1. Proton pump inhibitors (patients may switch to H2 blockers up to Day -7)
2. Inducers of P-gp (including, but not limited to, dexamethasone, morphine, ritonavir, saquinavir, tipranavir)
3. Moderate to potent inducers of CYP2B6, CYP2C8, or CYP3A4 (including, but not limited to, efavirenz, etavirine, modafinil, rifampin, St. John's Wort, carbamazepine, phenytoin) 19. History of taking any dose of amiodarone within 6 months (180 days) of Day 0

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2020-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Sulkowski, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital : The John G. Bartlett Specialty Practice, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sachithanandham J, Leep-Lazar J, Quinn J, Bowden K, Balasubramaniam P, Ward K, Ribeiro RM, Sulkowski MS, Balagopal A. Direct-Acting Antivirals Quickly Eradicate Hepatitis C Virus From the Liver in People With Human Immunodeficiency Virus but Do Not Fully Reverse Immune Activation. J Infect Dis. 2025 Jun 2;231(5):1299-1308. doi: 10.1093/infdis/jiae598. PMID 39656808
- [Derived] Sachithanandham J, Balagopal A, Leep-Lazar J, Quinn J, Bowden K, Ward K, Ribeiro RM, Sulkowski MS. Second-Phase Hepatitis C Plasma Viral Kinetics Directly Reflects Reduced Intrahepatic Burden of Hepatitis C Virus. J Infect Dis. 2023 Aug 11;228(3):311-320. doi: 10.1093/infdis/jiad025. PMID 36722133

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group A | Group B | Group C
Started | 5 | 5 | 5
Completed | 5 | 5 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Total
Number analyzed (Participants) | 5 | 5 | 5 | 15
Age, Continuous [Mean (Full Range); unit: years] | 50 [39 to 59] | 47 [28 to 60] | 54.6 [34 to 66] | 50.5 [28 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 7
  Male | 3 | 2 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 5 | 5 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 3 | 5 | 12
  White | 1 | 2 | 0 | 3
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: Total Number of HCV-infected Hepatocytes Measured in Liver Tissue Obtained by Liver Biopsy at Day 0 (Pre-treatment) and at Day 7 of Antiviral Therapy
Description: Estimate the total number of HCV-infected Hepatocytes (virus burden) for each participant between pre-treatment liver biopsy and post treatment liver biopsy samples using HCV Quantitative real time PCR.
  Comparison of total number of HCV-infected Hepatocytes (virus burden) were reported between HCV mono infection and co infection groups.
Time Frame: Pre-treatment, Day 7
Population: Overall number analyzed is the total hepatocytes analyzed in specific arms but numbers in rows represent only HCV positive Hepatocytes
Measure: Number; unit: Hepatocytes
Units Other Than Participants: Hepatocytes
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 5 | 5 | 5
Number analyzed (Hepatocytes) | 3220 | 3340 | 3463
Hepatocytes
  Participant 1 (Group A) Participant 1 (Group B) Participant 1 (Group C)pre trea: number analyzed (Participants) | 1 | 1 | 1
  Participant 1 (Group A) Participant 1 (Group B) Participant 1 (Group C)pre trea: number analyzed (Hepatocytes) | 247 | 265 | 335
  Participant 1 (Group A) Participant 1 (Group B) Participant 1 (Group C)pre trea | 45 | 16 | 290
  Participant 1 (Group A) Participant 1 (Group B) Participant 1 (Group C)pos trea: number analyzed (Participants) | 1 | 1 | 1
  Participant 1 (Group A) Participant 1 (Group B) Participant 1 (Group C)pos trea: number analyzed (Hepatocytes) | 351 | 345 | 347
  Participant 1 (Group A) Participant 1 (Group B) Participant 1 (Group C)pos trea | 2 | 5 | 7
  Participant 2 (Group A) Participant 2 (Group B) Participant 2 (Group C)pre trea: number analyzed (Participants) | 1 | 1 | 1
  Participant 2 (Group A) Participant 2 (Group B) Participant 2 (Group C)pre trea: number analyzed (Hepatocytes) | 326 | 349 | 358
  Participant 2 (Group A) Participant 2 (Group B) Participant 2 (Group C)pre trea | 53 | 11 | 33
  Participant 2 (Group A) Participant 2 (Group B) Participant 2 (Group C)pos trea: number analyzed (Participants) | 1 | 1 | 1
  Participant 2 (Group A) Participant 2 (Group B) Participant 2 (Group C)pos trea: number analyzed (Hepatocytes) | 342 | 350 | 353
  Participant 2 (Group A) Participant 2 (Group B) Participant 2 (Group C)pos trea | 0 | 1 | 3
  Participant 3 (Group A) Participant 3 (Group B) Participant 3 (Group C)pretreat: number analyzed (Participants) | 1 | 1 | 1
  Participant 3 (Group A) Participant 3 (Group B) Participant 3 (Group C)pretreat: number analyzed (Hepatocytes) | 334 | 359 | 355
  Participant 3 (Group A) Participant 3 (Group B) Participant 3 (Group C)pretreat | 18 | 212 | 216
  Participant 3 (Group A) Participant 3 (Group B) Participant 3 (Group C)postreat: number analyzed (Participants) | 1 | 1 | 1
  Participant 3 (Group A) Participant 3 (Group B) Participant 3 (Group C)postreat: number analyzed (Hepatocytes) | 339 | 352 | 346
  Participant 3 (Group A) Participant 3 (Group B) Participant 3 (Group C)postreat | 2 | 9 | 24
  Participant 4 (Group A) Participant 4 (Group B) Participant 4 (Group C)pre trea: number analyzed (Participants) | 1 | 1 | 1
  Participant 4 (Group A) Participant 4 (Group B) Participant 4 (Group C)pre trea: number analyzed (Hepatocytes) | 316 | 335 | 348
  Participant 4 (Group A) Participant 4 (Group B) Participant 4 (Group C)pre trea | 109 | 24 | 13
  Participant 4 (Group A) Participant 4 (Group B) Participant 4 (Group C)pos trea: number analyzed (Participants) | 1 | 1 | 1
  Participant 4 (Group A) Participant 4 (Group B) Participant 4 (Group C)pos trea: number analyzed (Hepatocytes) | 331 | 342 | 337
  Participant 4 (Group A) Participant 4 (Group B) Participant 4 (Group C)pos trea | 3 | 1 | 0
  Participant 5 (Group A) Participant 5 (Group B) Participant 5 (Group C)pretre: number analyzed (Participants) | 1 | 1 | 1
  Participant 5 (Group A) Participant 5 (Group B) Participant 5 (Group C)pretre: number analyzed (Hepatocytes) | 322 | 315 | 352
  Participant 5 (Group A) Participant 5 (Group B) Participant 5 (Group C)pretre | 126 | 4 | 74
  Participant 5 (Group A) Participant 5 (Group B) Participant 5 (Group C)postre: number analyzed (Participants) | 1 | 1 | 1
  Participant 5 (Group A) Participant 5 (Group B) Participant 5 (Group C)postre: number analyzed (Hepatocytes) | 312 | 328 | 332
  Participant 5 (Group A) Participant 5 (Group B) Participant 5 (Group C)postre | 18 | 1 | 12

2. Secondary Outcome: Reduction Over the First Week in Plasma HCV RNA
Description: During one week after treatment with direct-acting antivirals, the decline from the baseline plasma HCV RNA levels observed for each individual participant using HCV Quantitative real time PCR.
  The level of HCV RNA decline compared to those treated with Sofosbuvir/Velpatasvir (SOF/VEL) vs Sofosbuvir/Velpatasvir/Voxilaprevir (SOF/VEL/VOX) and between HCV mono infection and HIV/HCV co infection groups.
Time Frame: Pre-treatment, up to 1 week
Population: Decline plasma levels of HCV RNA from each participant obtained over the first week.
Measure: Median (Full Range); unit: IU/ml
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 5 | 5 | 5
IU/ml
  Participant 1 (Group A) Participant 1 (Group B) Participant 1 (Group C): number analyzed (Participants) | 1 | 1 | 1
  Participant 1 (Group A) Participant 1 (Group B) Participant 1 (Group C) | 631 [0 to 1945000] | 2240 [0 to 1760000] | 14817.5 [0 to 32700000]
  Participant 2 (Group A) Participant 2 (Group B) Participant 2 (Group C): number analyzed (Participants) | 1 | 1 | 1
  Participant 2 (Group A) Participant 2 (Group B) Participant 2 (Group C) | 217.75 [0 to 1080000] | 884.75 [0 to 478500] | 635.5 [0 to 1690000]
  Participant 3 (Group A) Participant 3 (Group B) Participant 3 (Group C): number analyzed (Participants) | 1 | 1 | 1
  Participant 3 (Group A) Participant 3 (Group B) Participant 3 (Group C) | 1029.75 [0 to 555500] | 1348500 [0 to 84300000] | 5327.5 [0 to 33050000]
  Participant 4 (Group A) Participant 4 (Group B) Participant 4 (Group C): number analyzed (Participants) | 1 | 1 | 1
  Participant 4 (Group A) Participant 4 (Group B) Participant 4 (Group C) | 6617.5 [0 to 14950000] | 551.5 [0 to 1020000] | 65075 [0 to 4675000]
  Participant 5 (Group A) Participant 5 (Group B) Participant 5 (Group C): number analyzed (Participants) | 1 | 1 | 1
  Participant 5 (Group A) Participant 5 (Group B) Participant 5 (Group C) | 2506.5 [0 to 4170000] | 627.5 [0 to 1680000] | 12992.5 [0 to 2990000]

3. Secondary Outcome: Total Number of HCV-infected Hepatocytes That Express Interferon-stimulated Genes (ISGs) Within the First Week of DAA Therapy Using Single Cell Laser Micro Dissection (scLCM).
Description: Total number of hepatocytes that express interferon-stimulated genes (ISGs) were estimated using Quantitative real time PCR for each participant on pre-treatment and post treatment liver biopsy samples.
  Comparison of total number of hepatocytes that express interferon-stimulated genes (ISGs) were reported between HCV mono infection and co infection groups.
Time Frame: Pre-treatment, up to 1 week
Population: Total number of hepatocytes that express interferon-stimulated genes (ISGs) between pre and post treatment
Measure: Number; unit: ISG positive hepatocytes
Units Other Than Participants: Hepatocytes
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 5 | 5 | 5
Number analyzed (Hepatocytes) | 904 | 912 | 904
ISG positive hepatocytes
  Participant 1 (Group A) Participant 1 (Group B) Participant 1 (Group C) Pre Treatment: number analyzed (Participants) | 1 | 1 | 1
  Participant 1 (Group A) Participant 1 (Group B) Participant 1 (Group C) Pre Treatment: number analyzed (Hepatocytes) | 88 | 96 | 96
  Participant 1 (Group A) Participant 1 (Group B) Participant 1 (Group C) Pre Treatment | 14 | 71 | 41
  Participant 1 (Group A) Participant 1 (Group B) Participant 1 (Group C) Post Treatment: number analyzed (Participants) | 1 | 1 | 1
  Participant 1 (Group A) Participant 1 (Group B) Participant 1 (Group C) Post Treatment: number analyzed (Hepatocytes) | 96 | 88 | 88
  Participant 1 (Group A) Participant 1 (Group B) Participant 1 (Group C) Post Treatment | 8 | 68 | 68
  Participant 2 (Group A) Participant 2 (Group B) Participant 2 (Group C) Pre Treatment: number analyzed (Participants) | 1 | 1 | 1
  Participant 2 (Group A) Participant 2 (Group B) Participant 2 (Group C) Pre Treatment: number analyzed (Hepatocytes) | 88 | 88 | 88
  Participant 2 (Group A) Participant 2 (Group B) Participant 2 (Group C) Pre Treatment | 57 | 36 | 39
  Participant 2 (Group A) Participant 2 (Group B) Participant 2 (Group C) Post Treatment: number analyzed (Participants) | 1 | 1 | 1
  Participant 2 (Group A) Participant 2 (Group B) Participant 2 (Group C) Post Treatment: number analyzed (Hepatocytes) | 96 | 88 | 88
  Participant 2 (Group A) Participant 2 (Group B) Participant 2 (Group C) Post Treatment | 62 | 24 | 40
  Participant 3 (Group A) Participant 3 (Group B) Participant 3 (Group C) Pre Treatment: number analyzed (Participants) | 1 | 1 | 1
  Participant 3 (Group A) Participant 3 (Group B) Participant 3 (Group C) Pre Treatment: number analyzed (Hepatocytes) | 88 | 96 | 88
  Participant 3 (Group A) Participant 3 (Group B) Participant 3 (Group C) Pre Treatment | 78 | 66 | 55
  Participant 3 (Group A) Participant 3 (Group B) Participant 3 (Group C) Post Treatment: number analyzed (Participants) | 1 | 1 | 1
  Participant 3 (Group A) Participant 3 (Group B) Participant 3 (Group C) Post Treatment: number analyzed (Hepatocytes) | 88 | 96 | 96
  Participant 3 (Group A) Participant 3 (Group B) Participant 3 (Group C) Post Treatment | 83 | 46 | 57
  Participant 4 (Group A) Participant 4 (Group B) Participant 4 (Group C) Pre Treatment: number analyzed (Participants) | 1 | 1 | 1
  Participant 4 (Group A) Participant 4 (Group B) Participant 4 (Group C) Pre Treatment: number analyzed (Hepatocytes) | 88 | 88 | 96
  Participant 4 (Group A) Participant 4 (Group B) Participant 4 (Group C) Pre Treatment | 71 | 49 | 36
  Participant 4 (Group A) Participant 4 (Group B) Participant 4 (Group C) Post Treatment: number analyzed (Participants) | 1 | 1 | 1
  Participant 4 (Group A) Participant 4 (Group B) Participant 4 (Group C) Post Treatment: number analyzed (Hepatocytes) | 96 | 88 | 88
  Participant 4 (Group A) Participant 4 (Group B) Participant 4 (Group C) Post Treatment | 71 | 27 | 63
  Participant 5 (Group A) Participant 5 (Group B) Participant 5 (Group C) Pre Treatment: number analyzed (Participants) | 1 | 1 | 1
  Participant 5 (Group A) Participant 5 (Group B) Participant 5 (Group C) Pre Treatment: number analyzed (Hepatocytes) | 88 | 88 | 88
  Participant 5 (Group A) Participant 5 (Group B) Participant 5 (Group C) Pre Treatment | 79 | 67 | 34
  Participant 5 (Group A) Participant 5 (Group B) Participant 5 (Group C) Post Treatment: number analyzed (Participants) | 1 | 1 | 1
  Participant 5 (Group A) Participant 5 (Group B) Participant 5 (Group C) Post Treatment: number analyzed (Hepatocytes) | 88 | 96 | 88
  Participant 5 (Group A) Participant 5 (Group B) Participant 5 (Group C) Post Treatment | 72 | 66 | 42

4. Secondary Outcome: Amount of HCV RNA Per Infected Hepatocyte Using Single Cell Laser Micro Dissection (scLCM) on Liver Biopsy Specimens, Obtained Just Prior to Treatment Initiation (Pre-treatment), and After the First Week of DAA Therapy.
Description: The HCV RNA levels (viral burden) from each infected hepatocytes were measured using Quantitative Real-Time Polymerase Chain Reaction (PCR) from each participants at pre-treatment and post-treatment.
  The level of HCV RNA (viral burden) decline were reported from intracellular hepatocytes and compared to those treated with Sofosbuvir/Velpatasvir (SOF/VEL) vs Sofosbuvir/Velpatasvir/Voxilaprevir (SOF/VEL/VOX) and between HCV mono infection and HIV/HCV co infection groups.
Time Frame: Pre-treatment, after first week
Population: Amount of HCV RNA levels from individual hepatocytes for each participant obtained at pre-treatment and post treatment.
Measure: Median (Full Range); unit: International unit (IU) per hepatocyte
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 5 | 5 | 5
International unit (IU) per hepatocyte
  Participant 1 (Group A) Participant 1 (Group B) Participant 1 (Group C) Pre treat: number analyzed (Participants) | 1 | 1 | 1
  Participant 1 (Group A) Participant 1 (Group B) Participant 1 (Group C) Pre treat | 8.61 [0.94 to 51.6] | 7.57 [0.1 to 41.1] | 32.7 [0.03 to 789]
  Participant 1 (Group A) Participant 1 (Group B) Participant 1 (Group C) Post treat: number analyzed (Participants) | 1 | 1 | 1
  Participant 1 (Group A) Participant 1 (Group B) Participant 1 (Group C) Post treat | 20.91 [10.47 to 29.7] | 2.83 [1.52 to 8.16] | 37.8 [3.39 to 274.8]
  Participant 2 (Group A) Participant 2 (Group B) Participant 2 (Group C)Pre treat: number analyzed (Participants) | 1 | 1 | 1
  Participant 2 (Group A) Participant 2 (Group B) Participant 2 (Group C)Pre treat | 19.74 [1.41 to 231.9] | 11.04 [5.94 to 54.6] | 18.36 [8.31 to 80.4]
  Participant 2 (Group A) Participant 2 (Group B) Participant 2 (Group C)Post treat: number analyzed (Participants) | 1 | 1 | 1
  Participant 2 (Group A) Participant 2 (Group B) Participant 2 (Group C)Post treat | 0 [0 to 0] | 12.93 [12.93 to 12.93] | 8.16 [2.89 to 17.16]
  Participant 3 (Group A) Participant 3 (Group B) Participant 3 (Group C)Pre treat: number analyzed (Participants) | 1 | 1 | 1
  Participant 3 (Group A) Participant 3 (Group B) Participant 3 (Group C)Pre treat | 10.35 [3.57 to 192.9] | 27.18 [1.37 to 336] | 30 [0.08 to 1584]
  Participant 3 (Group A) Participant 3 (Group B) Participant 3 (Group C)Post treat: number analyzed (Participants) | 1 | 1 | 1
  Participant 3 (Group A) Participant 3 (Group B) Participant 3 (Group C)Post treat | 14.76 [6.48 to 23] | 9.25 [3.21 to 47.1] | 15.72 [2.92 to 42]
  Participant 4 (Group A) Participant 4 (Group B) Participant 4 (Group C)Pre treat: number analyzed (Participants) | 1 | 1 | 1
  Participant 4 (Group A) Participant 4 (Group B) Participant 4 (Group C)Pre treat | 29.25 [1 to 187.2] | 3.45 [1 to 67.5] | 14.25 [1 to 72]
  Participant 4 (Group A) Participant 4 (Group B) Participant 4 (Group C)Post treat: number analyzed (Participants) | 1 | 1 | 1
  Participant 4 (Group A) Participant 4 (Group B) Participant 4 (Group C)Post treat | 9.15 [6.54 to 17.4] | 0 [0 to 0] | 0 [0 to 0]
  Participant 5 (Group A) Participant 5 (Group B) Participant 5 (Group C)Pre treat: number analyzed (Participants) | 1 | 1 | 1
  Participant 5 (Group A) Participant 5 (Group B) Participant 5 (Group C)Pre treat | 15.3 [0.15 to 738] | 2.36 [1.17 to 16.2] | 5.49 [0.008 to 33.9]
  Participant 5 (Group A) Participant 5 (Group B) Participant 5 (Group C)Post treat: number analyzed (Participants) | 1 | 1 | 1
  Participant 5 (Group A) Participant 5 (Group B) Participant 5 (Group C)Post treat | 14.55 [2 to 130.5] | 2.27 [2.27 to 2.27] | 4.09 [1.75 to 23.94]

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: adverse events were systematically assessed days 0-7, and week 2 and 4 study visits and as needed. Serious adverse events were systematically assessed at all follow-up visits and as needed.
Arm/Group | Group A | Group B | Group C
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 2/5 | 2/5 | 3/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=5) | Group B (N=5) | Group C (N=5)
Fatigue (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Flu-like symptoms (General disorders) | 0 (0) | 1 (1) | 0 (0)
Akathisia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) — One female participant became pregnant in the follow-up period of the study. While she was not exposed to the investigational agent during her pregnancy, this was reported to Gilead Sciences as a voluntary report.

LIMITATIONS AND CAVEATS:
This study is based on a relatively small sample of the liver

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-30): https://cdn.clinicaltrials.gov/large-docs/13/NCT02938013/Prot_SAP_000.pdf